CLINICAL TRIAL: NCT00384033
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Duloxetine-Referenced, Parallel-Group Study to Evaluate the Efficacy and Safety of 2 Fixed Doses (50mg, 100mg) of Desvenlafaxine Sustained-Release Tablets in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) In The Treatment Of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-335
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-02

CONDITIONS: Depressive Disorder, Major
Keywords: MDD; Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Desvenlafaxine succinate sustained-release 50 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
- Desvenlafaxine succinate sustained-release 100 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Duloxetine 60mg (Other): Active control to assess assay sensitivity
  Interventions: Drug: Duloxetine 60 mg/day

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR) — 50 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained-release 50 mg
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR) — 100 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained-release 100 mg
Drug: Placebo — Matching placebo tablets and capsules, once daily dosing for 8 weeks
  Arms: Placebo
Drug: Duloxetine 60 mg/day — 60 mg capsule, once daily dosing for 8 weeks
  Arms: Duloxetine 60mg

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of two doses of DVS SR (50 and 100 mg/day) in the treatment of adults with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of Major Depressive Disorder, single or recurrent episode, without psychotic features.
* Depressive symptoms for at least 30 days before the screening visit.
* Outpatient men and women at least 18 years of age.

Exclusion Criteria:

* Significant risk of suicide based on clinical judgment, including common suicidal thoughts and suicide having been considered as a possible solution even without specific plans or intent.
* Any unstable hepatic, renal, pulmonary, cardiovascular (including uncontrolled hypertension), ophthalmologic, neurologic, or any other medical condition that might confound the study or put the subject at greater risk during study participation.
* Current (within 12 months before baseline) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder; b) current (within 12 months before baseline) generalized anxiety disorder, panic disorder, or social anxiety disorder; c) presence (within 12 months before baseline) of a clinically important personality disorder as assessed during the psychiatric assessments.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Edwardsville, Illinois
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Okemos, Michigan
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Brown Deer, Wisconsin

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916
- [Derived] Tourian KA, Padmanabhan SK, Groark J, Brisard C, Farrington D. Desvenlafaxine 50 and 100 mg/d in the treatment of major depressive disorder: an 8-week, phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial and a post hoc pooled analysis of three studies. Clin Ther. 2009 Jun;31 Pt 1:1405-23. doi: 10.1016/j.clinthera.2009.07.006. PMID 19698901
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-335&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained%20Release%20%28DVS%20SR%29%20In%20The%20Treatment%20Of%20Major%20Depressive%20Disorder%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 27 September 2006 to 28 September 2007 in United States (US) only.
Pre-assignment Details: A total of 925 participants were screened for this study and 638 participants were randomized. The remaining 287 participants were not randomized due to screen failures.
Groups:
- Placebo: Placebo matched to desvenlafaxine succinate monohydrate sustained release (DVS SR) 50 milligram (mg) and 100 mg tablet and duloxetine 60 mg capsule daily until Day 56 (Week 8) or early termination (ET); then placebo matched to DVS SR 50 mg and 100 mg tablet and duloxetine 30 mg capsule for days 57-63 (Taper week).
- DVS SR 50 mg: DVS SR 50 mg tablet and placebo matched to DVS SR 100 mg tablet and duloxetine 60 mg capsule daily until Day 56 (Week 8) or ET; then placebo matched to DVS SR 50 mg and 100 mg tablet and duloxetine 30 mg capsule for days 57-63 (Taper week).
- DVS SR 100 mg: DVS SR 50 mg tablet and placebo matched to DVS SR 100 mg tablet and duloxetine 60 mg capsule daily for days 1-7; then DVS titrated up to 100 mg tablet, placebo matched to DVS SR 50 mg and duloxetine 60 mg capsule daily from days 8-56 (Week 8) or ET; then tapered to DVS SR 50 mg tablet and placebo matched to DVS SR 100 mg tablet and duloxetine 30 mg capsule for days 57-63 (Taper week).
- Duloxetine 60 mg: Duloxetine 60 mg capsule and placebo matched to DVS SR 50 mg and DVS SR 100 mg tablet daily until Day 56 (Week 8) or ET; then duloxetine 30 mg capsule and placebo matched to DVS SR 50 mg and 100 mg tablet for days 57-63 (Taper week).
Period: Overall Study
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Started | 164 | 155 | 160 | 159
Treated | 161 | 148 | 150 | 157
Completed | 123 | 120 | 117 | 119
Not Completed | 41 | 35 | 43 | 40
Not completed — Adverse Event | 10 | 8 | 11 | 20
Not completed — Failed to return | 1 | 3 | 2 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 12 | 7 | 7
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 5 | 6
Not completed — Withdrawal by Subject | 6 | 2 | 5 | 2
Not completed — Lack of Efficacy | 7 | 3 | 3 | 1
Not completed — Randomized but not treated | 3 | 7 | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 161 | 148 | 150 | 157 | 616
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.24 (12.74) | 40.67 (13.20) | 38.77 (12.07) | 38.94 (12.01) | 39.39 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 102 | 99 | 104 | 399
  Male | 67 | 46 | 51 | 53 | 217
Hamilton psychiatric scale for depression-17 item (HAM-D17) total score [Mean (Standard Deviation); unit: Units on a Scale] — HAM-D17: a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0 = none/absent and 4 = most severe, for a maximum total score of 50. N=160 for placebo treatment group.
  Units on a Scale | 23.86 (2.68) | 23.49 (2.52) | 23.49 (2.55) | 22.99 (2.45) | 23.46 (2.57)
Clinical global impressions scale-severity (CGI-S) score [Mean (Standard Deviation); unit: Units on a Scale] — CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill participants). Higher score = more affected. N=160 for placebo treatment group.
  Units on a Scale | 4.39 (0.54) | 4.29 (0.48) | 4.31 (0.49) | 4.28 (0.46) | 4.32 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HAM-D17 Total Score at Week 8 or Final On-therapy (FOT) Evaluation
Description: HAM-D17: a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0 = none/absent and 4 = most severe, for a maximum total score of 50.
Time Frame: Baseline and Week 8 or FOT
Population: Intent-to-treat (ITT) population included all randomized participants who had a baseline primary efficacy evaluation, had taken at least 1 dose of double-blind study medication, and had at least 1 primary efficacy evaluation after the first dose of double-blind study medication.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale | -8.68 (0.58) | -9.75 (0.60) | -10.5 (0.60) | -10.3 (0.60)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, HAM-D17 total score was evaluated using analysis of covariance (ANCOVA) with treatment and site as factors and baseline HAM-D17 score as the covariate; Test type: Superiority or Other; p = 0.198, ANCOVA — The analysis was done at a significance level of alpha = 0.05, 2-sided. Global F-test was used to adjust for multiplicity. If global F-test was significant at 0.05 level, pair wise analysis was interpreted without any further p-value adjustment; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [-0.60 to 2.70]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, HAM-D17 total score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D17 score as the covariate; Test type: Superiority or Other; p = 0.028, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.80, 95% CI 2-sided [0.20 to 3.40]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, HAM-D17 total score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D17 score as the covariate; Test type: Superiority or Other; p = 0.047, ANCOVA — The analysis was done at a significance level of alpha = 0.05, 2-sided, without any adjustments for multiple comparisons; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [0.00 to 3.40]

2. Secondary Outcome: Number of Participants With Categorical Scores on CGI-Improvement (CGI-I) Score at Week 8 or FOT Evaluation
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale relative to the baseline assessment. Higher score = more affected.
Time Frame: Week 8 or FOT
Population: ITT population included all randomized participants who had a baseline primary efficacy evaluation, had taken at least 1 dose of double-blind study medication, and had at least 1 primary efficacy evaluation after the first dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Participants
  1 = Very much improved | 31 | 27 | 45 | 45
  2 = Much improved | 32 | 38 | 37 | 35
  3 = Minimally improved | 35 | 47 | 28 | 37
  4 = No change | 57 | 34 | 37 | 37
  5 = Minimally worse | 5 | 2 | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, CGI-I was evaluated using Cochran-Mantel-Haenszel (CMH) test with treatment as a factor and controlling for center; Test type: Superiority or Other; p = 0.110, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, CGI-I was evaluated using CMH test with treatment as a factor and controlling for center; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, CGI-I was evaluated using CMH test with treatment as a factor and controlling for center; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]

3. Secondary Outcome: Change From Baseline in Mean CGI-S Score at Week 8 or FOT Evaluation
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill participants). Higher score = more affected.
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale | -1.10 (0.09) | -1.25 (0.10) | -1.44 (0.10) | -1.41 (0.10)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, CGI-S was evaluated using ANCOVA with treatment and site as factors and baseline CGI-S score as the covariate; Test type: Superiority or Other; p = 0.248, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.10 to 0.40]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, CGI-S was evaluated using ANCOVA with treatment and site as factors and baseline CGI-S score as the covariate; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [0.10 to 0.60]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, CGI-S was evaluated using ANCOVA with treatment and site as factors and baseline CGI-S score as the covariate; Test type: Superiority or Other; p = 0.026, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Median Difference (Final Values) = 0.30, 95% CI 2-sided [0.00 to 0.60]

4. Secondary Outcome: Change From Baseline in Montgomery and Asberg Depression Rating Scale (MADRS) Total Score at Week 8 or FOT Evaluation
Description: MADRS measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale
  Baseline | 31.10 (NA) — Standard error (SE) for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 30.10 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 30.70 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 30.80 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Change at Week 8 or FOT | -11.00 (0.82) | -12.70 (0.85) | -14.40 (0.84) | -14.40 (0.87)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, MADRS total score was evaluated using ANCOVA with treatment and site as factors and baseline MADRS score as the covariate; Test type: Superiority or Other; p = 0.149, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [-0.60 to 4.00]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, MADRS total score was evaluated using ANCOVA with treatment and site as factors and baseline MADRS score as the covariate; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.30, 95% CI 2-sided [1.10 to 5.60]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, MADRS total score was evaluated using ANCOVA with treatment and site as factors and baseline MADRS score as the covariate; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.40, 95% CI 2-sided [1.10 to 5.80]

5. Secondary Outcome: Change From Baseline in the Lassitude Item of the MADRS Scale at Week 8 or FOT Evaluation
Description: Lassitude item of MADRS represents a difficulty in getting started or slowness in initiating and performing everyday activities. It is rated on a scale of 0-6: 0 = hardly any difficulty in getting started/no sluggishness; 2 = difficulties in starting activities; 4 = difficulties in starting simple routine activities which are carried out with effort; 6 = complete lassitude/unable to do anything without help.
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale
  Baseline | 3.49 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 3.53 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 3.70 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 3.50 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Change at Week 8 or FOT | -1.27 (0.12) | -1.39 (0.13) | -1.54 (0.13) | -1.26 (0.12)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, lassitude item of the MADRS score was evaluated using ANCOVA with treatment and site as factors and baseline lassitude item of the MADRS score as the covariate; Test type: Superiority or Other; p = 0.473, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.22 to 0.46]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, lassitude item of the MADRS score was evaluated using ANCOVA with treatment and site as factors and baseline lassitude item of the MADRS score as the covariate; Test type: Superiority or Other; p = 0.119, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.07 to 0.61]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, lassitude item of the MADRS score was evaluated using ANCOVA with treatment and site as factors and baseline lassitude item of the MADRS score as the covariate; Test type: Superiority or Other; p = 0.710, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.27 to 0.40]

6. Secondary Outcome: Change From Baseline in HAM-D6 Total Score at Week 8 or FOT Evaluation
Description: HAM-D6: a standardized, clinician-administered rating scale that assesses 6 items characteristically associated with major depression and is a subset of HAM-D17. HAM-D6 score ranges from 0-22. The scale uses HAM-D17 items: 1, 2, 7, 8, 10 and 13. Item 13 is scored 0-2 (0=none and 2=severe) and all others are scored 0-4 (0=none/absent and 4=most severe).
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale
  Baseline | 13.00 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 12.80 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 12.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 12.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Change at Week 8 or FOT | -4.82 (0.33) | -5.41 (0.35) | -6.15 (0.34) | -5.91 (0.36)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, HAM-D6 score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D6 score as the covariate; Test type: Superiority or Other; p = 0.215, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-0.30 to 1.50]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, HAM-D6 score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D6 score as the covariate; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [0.40 to 2.30]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, HAM-D6 score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D6 score as the covariate; Test type: Superiority or Other; p = 0.024, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.20 to 2.10]

7. Secondary Outcome: Change From Baseline in the HAM-D Energy Subscale Score at Week 8 or FOT Evaluation
Description: HAM-D energy subscale is a subset of the HAM-D17 that assesses 4 items associated with major depression. The scale uses HAM- D17 items 1, 7, 8 and 14. Item 14 is scored 0 to 2 (0=none/absent to 2=most severe) and all others are scored 0 to 4 (0=none/absent to 4=most severe).
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale
  Baseline | 8.38 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 8.43 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 8.51 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 8.38 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Change at Week 8 or FOT | -3.13 (0.23) | -3.66 (0.23) | -3.92 (0.23) | -3.80 (0.24)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, HAM-D energy subscale score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D energy score as the covariate; Test type: Superiority or Other; p = 0.100, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.10 to 1.17]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, HAM-D energy subscale score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D energy score as the covariate; Test type: Superiority or Other; p = 0.014, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [0.16 to 1.42]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, HAM-D energy subscale score was evaluated using ANCOVA with treatment and site as factors and baseline HAM-D energy score as the covariate; Test type: Superiority or Other; p = 0.032, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.06 to 1.38]

8. Secondary Outcome: Change From Baseline in Covi Anxiety Scale at Week 8 or FOT Evaluation
Description: COVI anxiety scale measures the severity of anxiety symptoms on 3 items: verbal report, behavior and somatic complaints. Each dimension is assessed using a 5-point scale: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = considerably, to 5 = Very much. Worst value is 15 and best value is 3.
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
Units on a Scale
  Baseline | 6.50 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 6.30 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 6.30 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 6.30 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Change at Week 8 or FOT | -1.02 (0.12) | -1.15 (0.13) | -1.35 (0.13) | -1.47 (0.13)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, Covi anxiety scale was evaluated using ANCOVA with treatment and site as factors and baseline Covi anxiety score as the covariate; Test type: Superiority or Other; p = 0.445, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.20 to 0.50]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, Covi anxiety scale was evaluated using ANCOVA with treatment and site as factors and baseline Covi anxiety score as the covariate; Test type: Superiority or Other; p = 0.056, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.00 to 0.70]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, Covi anxiety scale was evaluated using ANCOVA with treatment and site as factors and baseline Covi anxiety score as the covariate; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Median Difference (Final Values) = 0.50, 95% CI 2-sided [0.10 to 0.90]

9. Secondary Outcome: Change From Baseline in Visual Analog Scale-Pain Intensity (VAS-PI) Overall and Subcomponent Score at Week 8 or FOT Evaluation
Description: VAS-PI scale assesses intensity of back pain, chest pain, arms, legs or joint pain as well as overall pain intensity where 100 mm line (VAS) is marked by participant and intensity of pain ranges from 0 millimetre (mm) = no pain to 100 mm = worst possible pain. There were separate 0 to 100 mm VAS lines for each subcomponent of VAS-PI.
Time Frame: Baseline and Week 8 or FOT
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Number analyzed (Participants) | 160 | 148 | 150 | 157
mm
  Overall pain (Baseline) | 26.30 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 30.80 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 25.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 26.10 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Stomach pain (Baseline) | 16.70 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 19.40 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 17.00 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 14.00 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Back pain (Baseline) | 25.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 32.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 28.30 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 25.50 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Chest pain (Baseline) | 9.40 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 10.90 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 10.40 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 6.60 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Arms, legs or joint pain (Baseline) | 25.80 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 29.10 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 28.70 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison. | 22.40 (NA) — SE for baseline was not obtained for secondary variables as the focus was on adjusting for baseline, not on baseline comparison.
  Overall pain (Change at Week 8 or FOT) | -5.61 (1.57) | -9.08 (1.64) | -10.30 (1.63) | -8.84 (1.74)
  Stomach pain (Change at Week 8 or FOT) | -1.86 (1.62) | -4.98 (1.69) | -6.42 (1.68) | -4.38 (1.58)
  Back pain (Change at Week 8 or FOT) | -7.04 (1.67) | -10.70 (1.74) | -12.80 (1.73) | -9.33 (1.83)
  Chest pain (Change at Week 8 or FOT) | -1.95 (1.12) | -3.34 (1.17) | -3.90 (1.16) | -1.67 (1.21)
  Arms, legs or joint pain (Change at Week 8 or FOT) | -6.99 (1.70) | -8.98 (1.76) | -11.90 (1.76) | -8.35 (1.64)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, overall VAS-PI score was evaluated using ANCOVA with treatment and site as factors and baseline VAS-PI score as the covariate; Test type: Superiority or Other; p = 0.124, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.50, 95% CI 2-sided [-0.90 to 7.90]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, overall VAS-PI score was evaluated using ANCOVA with treatment and site as factors and baseline VAS-PI score as the covariate; Test type: Superiority or Other; p = 0.035, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [0.30 to 9.10]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, overall VAS-PI score was evaluated using ANCOVA with treatment and site as factors and baseline VAS-PI score as the covariate; Test type: Superiority or Other; p = 0.093, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Median Difference (Final Values) = 4.10, 95% CI 2-sided [-0.70 to 8.80]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, stomach pain score was evaluated using ANCOVA with treatment and site as factors and baseline stomach pain score as the covariate; Test type: Superiority or Other; p = 0.177, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.10, 95% CI 2-sided [-1.40 to 7.70]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, stomach pain score was evaluated using ANCOVA with treatment and site as factors and baseline stomach pain score as the covariate; Test type: Superiority or Other; p = 0.048, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 4.60, 95% CI 2-sided [0.10 to 9.10]
Statistical Analysis 6: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, stomach pain score was evaluated using ANCOVA with treatment and site as factors and baseline stomach pain score as the covariate; Test type: Superiority or Other; p = 0.088, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.80, 95% CI 2-sided [-0.50 to 8.10]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, back pain score was evaluated using ANCOVA with treatment and site as factors and baseline back pain score as the covariate; Test type: Superiority or Other; p = 0.122, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.70, 95% CI 2-sided [-1.00 to 8.40]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, back pain score was evaluated using ANCOVA with treatment and site as factors and baseline back pain score as the covariate; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 5.80, 95% CI 2-sided [1.10 to 10.50]
Statistical Analysis 9: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, back pain score was evaluated using ANCOVA with treatment and site as factors and baseline back pain score as the covariate; Test type: Superiority or Other; p = 0.103, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 4.20, 95% CI 2-sided [-0.80 to 9.20]
Statistical Analysis 10: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, chest pain score was evaluated using ANCOVA with treatment and site as factors and baseline chest pain score as the covariate; Test type: Superiority or Other; p = 0.384, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-1.70 to 4.50]
Statistical Analysis 11: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, chest pain score was evaluated using ANCOVA with treatment and site as factors and baseline chest pain score as the covariate; Test type: Superiority or Other; p = 0.221, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 2.00, 95% CI 2-sided [-1.20 to 5.10]
Statistical Analysis 12: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, chest pain score was evaluated using ANCOVA with treatment and site as factors and baseline chest pain score as the covariate; Test type: Superiority or Other; p = 0.411, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-1.90 to 4.70]
Statistical Analysis 13: Comparison: Placebo vs DVS SR 50 mg; For DVS SR 50 mg, arms, legs, joint pain score was evaluated using ANCOVA with treatment and site as factors and baseline arms, legs, pain score as the covariate; Test type: Superiority or Other; p = 0.412, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 2.00, 95% CI 2-sided [-2.80 to 6.70]
Statistical Analysis 14: Comparison: Placebo vs DVS SR 100 mg; For DVS SR 100 mg, arms, legs, joint pain score was evaluated using ANCOVA with treatment and site as factors and baseline arms, legs, pain score as the covariate; Test type: Superiority or Other; p = 0.042, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 4.90, 95% CI 2-sided [0.20 to 9.60]
Statistical Analysis 15: Comparison: Placebo vs Duloxetine 60 mg; For Duloxetine 60 mg, arms, legs, joint pain score was evaluated using ANCOVA with treatment and site as factors and baseline arms, legs, pain score as the covariate; Test type: Superiority or Other; p = 0.155, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 3.30, 95% CI 2-sided [-1.20 to 7.80]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 2/161 | 2/148 | 2/150 | 1/157
Other Adverse Events (participants affected / at risk) | 129/161 | 134/148 | 134/150 | 141/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | DVS SR 50 mg (N=148) | DVS SR 100 mg (N=150) | Duloxetine 60 mg (N=157)
Accidental injury (General disorders) | 1 | 1 | 0 | 0
Suicide attempt (General disorders) | 0 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Menorrhagia (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | DVS SR 50 mg (N=148) | DVS SR 100 mg (N=150) | Duloxetine 60 mg (N=157)
Abdominal pain (General disorders) | 12 | 8 | 8 | 15
Asthenia (General disorders) | 9 | 15 | 19 | 21
Back pain (General disorders) | 10 | 3 | 0 | 5
Flu syndrome (General disorders) | 8 | 7 | 12 | 5
Headache (General disorders) | 38 | 27 | 28 | 30
Infection (General disorders) | 7 | 10 | 15 | 6
Pain (General disorders) | 9 | 3 | 4 | 4
Withdrawal syndrome (General disorders) | 24 | 42 | 42 | 49
Anorexia (Gastrointestinal disorders) | 7 | 14 | 14 | 29
Constipation (Gastrointestinal disorders) | 5 | 9 | 10 | 17
Diarrhea (Gastrointestinal disorders) | 22 | 18 | 24 | 26
Dry mouth (Gastrointestinal disorders) | 25 | 26 | 31 | 33
Dyspepsia (Gastrointestinal disorders) | 9 | 8 | 10 | 7
Nausea (Gastrointestinal disorders) | 22 | 36 | 40 | 52
Vomitting (Gastrointestinal disorders) | 4 | 3 | 11 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 6 | 5
Abnormal dreams (Nervous system disorders) | 3 | 5 | 5 | 12
Anxiety (Nervous system disorders) | 11 | 4 | 2 | 4
Dizziness (Nervous system disorders) | 15 | 15 | 26 | 27
Insomnia (Nervous system disorders) | 9 | 23 | 28 | 37
Somnolence (Nervous system disorders) | 12 | 16 | 18 | 33
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 20 | 24 | 20 | 25
Sweating (Skin and subcutaneous tissue disorders) | 4 | 9 | 9 | 19
Abnormal vision (General disorders) | 2 | 8 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.